CLINICAL TRIAL: NCT02626234
Title: A Phase I, Multicenter, Open-label, Single-sequence Drug-drug Interaction Study to Assess the Effect of INC280 on the Pharmacokinetics of Digoxin and Rosuvastatin in Patients With cMET-dysregulated Advanced Solid Tumors
Brief Title: A Drug-drug Interaction (DDI) Study to Assess the Effect of INC280 on the Pharmacokinetics of Digoxin and Rosuvastatin in Patients With cMET-dysregulated Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC280A2105
Record Dates: First submitted 2015-10-13; First posted 2015-12-10 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-07

CONDITIONS: cMET-dysregulated Advanced Solid Tumors
Keywords: cMET, INC280, rosuvastatin, digoxin
MeSH Terms: interventions — capmatinib; Digoxin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INC280 (Experimental)
  Interventions: Drug: INC280; Drug: digoxin; Drug: rosuvastatin

INTERVENTIONS:
Drug: INC280
Drug: digoxin
Drug: rosuvastatin

SUMMARY:
the study aim to assess the effect of INC280 on the pharmacokinetics of digoxin and rosuvastatin in patients with cMET-dysregulated advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

Patients must have:

* advanced solid tumors and have confirmed cMET dysregulation
* at least one measurable lesion as defined by RECIST 1.1.
* recovered from all toxicities related to prior anti-cancer therapies
* adequate organ function
* ECOG performance status (PS) of 0 or 1

Exclusion Criteria:

Patients must not have:

* known hypersensitivity to any of the excipients of INC280
* prior treatment with cMET or HGF-targeting inhibitor
* known hypersensitivity to digoxin or rosuvastatin or its excipients
* symptomatic central nervous system (CNS) metastases who are neurologically unstable
* presence or history of carcinomatous meningitis
* history of another primary malignancy that is currently clinically significant or currently requires active intervention
* Clinically significant, uncontrolled heart diseases, including QTcF ≥ 450 msec (male patients), ≥ 460 msec (female patients) on the screening ECG
* Thoracic radiotherapy to lung fields ≤ 4 weeks prior to starting INC280
* Major surgery within 4 weeks prior to starting INC280
* Patients receiving unstable or increasing doses of corticosteroids.
* Impairment of GI function or GI disease that may significantly alter the absorption of INC280
* Patients who have received, or are expected to receive digoxin or rosuvastatin within 21 days prior to the beginning of the DDI phase (Day 1) and for the duration of the DDI phase.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
AUClast of digoxin and rosuvastatin | Up to 240 hours post digoxin and rosuvastatin dose
  digoxin and rosuvastatin pharmacokinetics parameters
AUCinf of digoxin and rosuvastatin | Up to 240 hours post digoxin and rosuvastatin dose
  digoxin and rosuvastatin pharmacokinetics parameters
Lambda_z of digoxin and rosuvastatin | Up to 240 hours post digoxin and rosuvastatin dose
  digoxin and rosuvastatin pharmacokinetics parameters
Cmax of digoxin and rosuvastatin | Up to 240 hours post digoxin and rosuvastatin dose
  digoxin and rosuvastatin pharmacokinetics parameters
Tmax of digoxin and rosuvastatin | Up to 240 hours post digoxin and rosuvastatin dose
  digoxin and rosuvastatin pharmacokinetics parameters
T1/2 of digoxin and rosuvastatin | Up to 240 hours post digoxin and rosuvastatin dose
  digoxin and rosuvastatin pharmacokinetics parameters
CL/F of digoxin and rosuvastatin | Up to 240 hours post digoxin and rosuvastatin dose
  digoxin and rosuvastatin pharmacokinetics parameters
Vz/F of digoxin and rosuvastatin | Up to 240 hours post digoxin and rosuvastatin dose
  digoxin and rosuvastatin pharmacokinetics parameters

SECONDARY OUTCOMES:
Adverse events based on the CTCAE v4.03 grade (severity) and other safety data (e.g.,ECG, vital signs, laboratory results) | From consent to 30 days post last dose
  To assess safety and tolerability of INC280 in patients with cMET-dysregulated advanced solid tumors
Overall response rate of patients treated with INC280 | Up to 12 months
  Overall response rate is defined as Complete Response and Partial Response calculated per RECIST 1.1, per investigator assessment from Day 1 until date of progression or death whichever comes first
Disease control rate of patients treated with INC280 | Up to 12 months
  Disease control rate is defined as calculated as the proportion of patients with best overall response of Complete Response, Partial Response, or Stable Disease calculated per RECIST 1.1, per investigator assessment from Day 1 until date of progression or death whichever comes first
Concentration of INC280 during DDI phase | Day 22, Cycle 2 Day 1
  INC280 concentrations collected on Day 22 during DDI phase and Cycle 2 Day 1 during post DDI phase along with a listing of individual values.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- United States (2):
  - Emory University School of Medicine/Winship Cancer Institute Phase 1 Working Group, Atlanta, Georgia
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Edegem, Antwerpen, Belgium
- Novartis Investigative Site, Brno, Czechia
- Greece (2):
  - Novartis Investigative Site, Ioannina, GR
  - Novartis Investigative Site, Athens
- Italy (4):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Candiolo, TO
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Madrid, Spain
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CINC280A2105 can be found Novartis Clinical trials results website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17087